CLINICAL TRIAL: NCT06147180
Title: Comparison of Long-term Survival and Quality of Life After Minimally Invasive Esophagectomy Versus Open Esophagectomy for Esophageal Cancer: a Retrospective Cohort Study
Brief Title: Comparison of Long-term Survival and Quality of Life After Minimally Invasive Esophagectomy Versus Open Esophagectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: MR-37-23-034233
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-10

CONDITIONS: Esophagus Cancer; Esophagectomy; Quality of Life; Survival
Keywords: esophagus Cancer; invasive esophagectomy; open esophagectomy; long-term survival; quality of life
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally invasive esophageal cancer resection group: Surgical Procedures: minimally invasive esophagectomy
- Open esophageal cancer resection group: Surgical Procedures: open esophagectomy

SUMMARY:
To analyze and compare the long-term recurrence-free survival rate, overall survival rate and quality of survival after minimally invasive esophagectomy and open esophagectomy, and to conduct subgroup analysis according to the type of esophageal cancer and pathological stage, etc., and to explore more deeply the differences between minimally invasive esophagectomy and open esophagectomy in terms of the benefits for different types of patients, so as to provide reference for the selection of the clinical surgical methods. We will also use the available data to analyze the influence of other factors on patients' long-term survival after surgery.

DETAILED DESCRIPTION:
1. Purpose of the study To study the differences in long-term disease-free survival rate and overall survival rate after minimally invasive esophagectomy and open esophagectomy, as well as postoperative quality of life, and to prove whether the choice of surgical modality has an impact on the postoperative long-term survival of esophageal cancer patients, and to explore the target population that can benefit more from minimally invasive esophagectomy compared with open esophagectomy, so as to provide a The study will also explore the target population that can benefit more from minimally invasive esophagectomy than open esophagectomy, so as to provide a certain reference value for the selection of surgical methods in clinics. To analyze the impact of other baseline data on patients' long-term survival and quality of life after surgery using the available data.
2. Content of the study To retrieve the electronic medical records of patients who had undergone esophageal cancer resection at the Department of Thoracic Surgery, Qilu Hospital, Shandong University, between 2013 and 2021, to collect their baseline data, and to classify patients into minimally invasive surgery and open surgery groups according to surgical modalities, and to match the propensity scores of patients in the two groups on the important baseline data, and to collect the postoperative recurrence of metastasis, survival, and the quality of life of the patients through the follow up visits To compare the long-term recurrence-free survival rate, overall survival rate and quality of life between the two groups, and to analyze the subgroups according to the type of esophageal cancer, pathological stage, and whether neoadjuvant therapy was performed, so as to explore more deeply the differences between minimally invasive esophagectomy and open esophagectomy in terms of postoperative long-term survival for patients with different types of esophageal cancers. And to analyze the influence of other baseline information on patients' postoperative long-term survival and quality of life.
3. Observed Indicators The main outcomes observed in this study were disease-free survival and overall survival after surgery.Survival was calculated: if the patient survived from the date of surgery to the date of follow-up, the survival period was from the date of surgery to the date of follow-up, and if the patient died between the date of surgery and the date of follow-up, the survival period was from the date of surgery to the date of death. Calculation of disease-free survival: from the date of surgery to the date of the first detection of recurrent metastatic disease between the date of surgery and the date of follow-up; the criterion for recurrence is the presence of metastases to other organs or lymph nodes after surgery confirmed by histology or imaging. Observation time: the patient's time from the first postoperative date to 5 full years postoperatively was taken as the observation time. Follow-up outcome: patient's death, loss to follow-up, or patient's survival at 5 full years postoperatively from the first postoperative date to 5 full years postoperatively were considered as the primary observation outcomes. Since the patients in this study were from patients who had undergone esophagectomy for esophageal cancer at the Department of Thoracic Surgery, Qilu Hospital, Shandong University, during the period 2013-2021, the follow-up period was set at 3 years from the date of ethical approval - 3 years after the ethical approval was granted, which would allow all patients to reach the observation period of 5 years, and for cancer patients, the 3 and 5 year survival rates are very important prognostic data.
4. Data collection Collection of patients' baseline data: baseline data of patients who had undergone esophagectomy for esophageal cancer at the Department of Thoracic Surgery, Qilu Hospital, Shandong University, and were successfully discharged from the hospital during the period from 2013 to 2021 were collected through the electronic medical record system, including, but not limited to, hospitalization number, name, gender, age, occupation, marital status, contact phone number, underlying disease, history of smoking and alcohol consumption, family history, PS score, body weight (kg), height (m ), ASA score, tumor site, date of surgery, duration of surgery (min), mode of surgery, intraoperative bleeding (ml), duration of surgery (min), blood routine, blood biochemistry, blood type, pathological results, lung function, postoperative course, and surgical complications. Collection of patients' postoperative survival data: follow-up to collect patients' postoperative survival data information, including, whether they were alive at the time of the follow-up date, the specific date of death, whether they died due to this disease, whether they had recurrent metastasis, the time of the first recurrent metastasis, and the information on the quality of postoperative survival, which was obtained according to the EORTC QLQ-OES18 quality of life questionnaire.
5. Statistical analysis For the baseline data collected from patients, it was initially planned to use propensity score matching, with the minimally invasive surgery group and the open surgery group in a 1:1 ratio, so that the data of the two groups would be consistent in terms of baseline data; after obtaining the survival data of the patients in the postoperative period, the comparison of the continuous variables was performed using the Wilcoxon test/Mann Whitney U test or Student t-test, and the categorical variables were analyzed using the Pearson chi-square test or Fisher exact test. Categorical variables were reported as frequencies, percentages, and P values, and continuous variables were reported as means, ranges, and P values. The long-term recurrence-free survival and overall survival rates of the two groups and their 95% CIs were analyzed, and the hazard ratios of recurrence-free survival and overall survival and the differences between recurrence-free survival and overall survival were compared to see whether the differences were statistically significant; if the differences in the survival rates were statistically significant, there was a certain relationship between the long-term survival of esophageal cancer and the surgical modality, and if the differences were not statistically significant, it indicated that the two surgical In subgroup analysis, the long-term recurrence-free survival rate and overall survival rate and their 95% CIs were calculated for squamous carcinoma, adenocarcinoma, other malignant tumors, and different pathological stage subgroups, and the hazard ratios of the recurrence-free survival rate and overall survival rate and the differences between the recurrence-free survival rate and overall survival rate of the two groups were compared between the subgroups to see whether the differences were statistically significant or not, the difference was statistically significant for subgroups with statistically significant differences, indicating that there was a certain relationship between postoperative survival and surgery. statistically significant subgroups suggests that the choice of surgical modality can benefit patients with that characteristic, and thus there is a tendency to choose a more beneficial surgical modality for patients in clinical work. On the other hand, the EORTC QLQ-OES18 quality of life questionnaire classified the outcomes into 10 domains such as dysphagia, and by collecting information on the quality of life of surviving patients, we analyzed and compared whether there were differences in the quality of life of the two groups of patients in the different functional domains, so as to compare whether there was any effect of surgical modality on the quality of life of the patients in the postoperative period. Utilizing the available information, other factors were explored to find out whether there was any influence of other factors on postoperative survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had undergone esophageal cancer resection at the Department of Thoracic Surgery, Qilu Hospital, Shandong University, between 2013 and 2021, with pathology results confirming esophageal squamous carcinoma, adenocarcinoma, or other malignant tumors.
2. The surgery was successfully completed, the patient was safely discharged from the hospital, the postoperative follow-up was successful, and if the follow-up patient died, his or her death was due to natural causes.

Exclusion Criteria:

Perioperative patient deaths, pathologic findings other than those listed above, loss of visits, and postoperative unnatural deaths.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had undergone esophageal cancer resection at the Department of Thoracic Surgery, Qilu Hospital, Shandong University, between 2013 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1474 (Estimated)
Dates: Start 2023-11-27 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Survival Information | From enrollment to 5 years after surgery
  Dead or alive 5 years after surgery
score of Quality of life | From enrollment to 5 years after surgery
  Measured with EORTC QLQ-OES18 Quality of Life Questionnaire

SECONDARY OUTCOMES:
Recurrence or metastasis | From enrollment to 5 years after surgery
  Imaging, lab results

CONTACTS AND LOCATIONS:
Overall Officials: Hui Tian, Doctor, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Z, Liu C, Liu Y, Yao S, Xu B, Dong G. Comparisons between minimally invasive and open esophagectomy for esophageal cancer with cervical anastomosis: a retrospective study. J Cardiothorac Surg. 2020 Jun 8;15(1):128. doi: 10.1186/s13019-020-01182-3. PMID 32513211
- [Background] Zheng Y, Li Y, Liu X, Sun H, Shen S, Ba Y, Wang Z, Liu S, Xing W. Minimally Invasive Versus Open McKeown for Patients with Esophageal Cancer: A Retrospective Study. Ann Surg Oncol. 2021 Oct;28(11):6329-6336. doi: 10.1245/s10434-021-10105-y. Epub 2021 May 13. PMID 33987755
- [Background] Ising MS, Smith SA, Trivedi JR, Martin RCG, Phillips P, Van Berkel V, Fox MP. Minimally Invasive Esophagectomy Is Associated with Superior Survival Compared to Open Surgery. Am Surg. 2023 May;89(5):1833-1843. doi: 10.1177/00031348221078962. Epub 2022 Mar 23. PMID 35317621
- [Background] Chen HS, Lin CH, Wu SC, Wang BY. Comparing survival between neoadjuvant chemoradiotherapy followed by open or thoracoscopic oesophagectomy in patients with oesophageal squamous cell carcinoma. Eur J Cardiothorac Surg. 2022 Jul 11;62(2):ezac114. doi: 10.1093/ejcts/ezac114. PMID 35303068
- [Background] van der Sluis PC, van der Horst S, May AM, Schippers C, Brosens LAA, Joore HCA, Kroese CC, Haj Mohammad N, Mook S, Vleggaar FP, Borel Rinkes IHM, Ruurda JP, van Hillegersberg R. Robot-assisted Minimally Invasive Thoracolaparoscopic Esophagectomy Versus Open Transthoracic Esophagectomy for Resectable Esophageal Cancer: A Randomized Controlled Trial. Ann Surg. 2019 Apr;269(4):621-630. doi: 10.1097/SLA.0000000000003031. PMID 30308612
- [Background] Knitter S, Andreou A, Hofmann T, Chopra S, Denecke C, Thuss-Patience PC, Kroll D, Bahra M, Schmelzle M, Pratschke J, Biebl M. Minimally Invasive Versus Open Ivor-Lewis Esophagectomy for Esophageal Cancer or Cancer of the Gastroesophageal Junction: Comparison of Postoperative Outcomes and Long-term Survival Using Propensity Score Matching Analysis. Anticancer Res. 2021 Jul;41(7):3499-3510. doi: 10.21873/anticanres.15137. PMID 34230145
- [Background] Gottlieb-Vedi E, Kauppila JH, Mattsson F, Lindblad M, Nilsson M, Lagergren P, Rouvelas I, Lagergren J; FINEGO group. Long-term Survival in Esophageal Cancer After Minimally Invasive Esophagectomy Compared to Open Esophagectomy. Ann Surg. 2022 Dec 1;276(6):e744-e748. doi: 10.1097/SLA.0000000000004645. Epub 2021 Jan 20. PMID 33480612
- [Background] Giulini L, Dubecz A. Minimally invasive versus open oesophagectomy for cancer: propensity score analysis improves results' reliability but matching criteria need to be selected accurately. Eur J Cardiothorac Surg. 2022 Jul 11;62(2):ezac192. doi: 10.1093/ejcts/ezac192. No abstract available. PMID 35349668